CLINICAL TRIAL: NCT07375173
Title: Oxygen Reserve Index-Guided FiO₂ Titration in Prone Spine Surgery: Impact on Postoperative Atelectasis Assessed by Lung Ultrasound
Brief Title: ORI-Guided FiO₂ Titration in Prone Spine Surgery: Impact on Postoperative Atelectasis Assessed by Lung Ultrasound
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Sıla Soytaş, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AEŞH-EK-2025-301
Record Dates: First submitted 2025-11-19; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Atelectases, Postoperative Pulmonary; Prone Position; Spine Surgery; Lung Ultrasound; Oxygen Reserve Index
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1-ORI-Guided FiO₂ Titration Group (Active Comparator): Patients will receive 80% FiO₂ for 3 minutes before induction. After intubation, FiO₂ will be set to 50% and titrated to keep the Oxygen Reserve Index (ORI) between 0.00-0.05 using the Masimo Rad-97. If ORI ≥0.05 for ≥5 min, FiO₂ will be reduced by 0.05; if ORI stays within 0-0.05 for ≥5 min, FiO₂ will be maintained; if ORI = 0 with SpO₂ <95%, FiO₂ will be increased by 0.05. The target PaO₂ is 80-120 mmHg. PEEP will be fixed at 5 cmH₂O, and a standard recruitment maneuver will be applied at surgery start. The protocol continues throughout the operation. Only noninvasive methods (ORI, LUS, spirometry) will be used. Both groups will have preoperative LUS and spirometry. Postoperative LUS will be repeated at 30 minutes and spirometry at 24 hours for comparative assessment.
  Interventions: Procedure: Titrated Oxygen
- Group 2- Fixed FiO₂ (Active Comparator): Patients will undergo preoxygenation with 80% FiO₂ for 3 minutes prior to induction. After endotracheal intubation, FiO₂ will be maintained at 50% and continued unchanged throughout the surgical procedure. Positive end-expiratory pressure (PEEP) will be set at 5 cmH₂O, and a standard alveolar recruitment maneuver will be applied to all patients at the beginning of surgery.
  The intervention will be continued throughout the surgical procedure. Only noninvasive monitoring (ORI measurement), lung ultrasonography (LUS), and spirometry will be performed in this study. In both groups, preoperative spirometry and lung ultrasonography will be conducted. Postoperatively, lung ultrasonography will be repeated at the 30th minute, and spirometry will be repeated at the 24th hour to allow for comparative analysis.
  Interventions: Procedure: Fixed oxygen

INTERVENTIONS:
Procedure: Titrated Oxygen — This intervention is distinguished by the use of real-time Oxygen Reserve Index (ORI) monitoring to guide individualized intraoperative FiO₂ titration. Unlike fixed-FiO₂ strategies commonly used in anesthesia practice, this protocol continuously adjusts FiO₂ based on ORI values measured with the Masimo Rad-97 device. FiO₂ is increased or decreased in increments of 0.05 according to predefined ORI thresholds to maintain patients within a targeted normoxemic range. The intervention is entirely noninvasive and integrates standardized lung ultrasound (LUS) assessments and spirometry to evaluate postoperative aeration loss and respiratory function. This dynamic, physiology-based oxygen management approach differentiates the intervention from routine fixed-oxygen administration used in other clinical studies.
  Other Names: Oxygen Reserve Index-Guided Oxygen Titration
  Arms: Group 1-ORI-Guided FiO₂ Titration Group
Procedure: Fixed oxygen — This intervention uses a standard, non-individualized oxygen administration approach in which FiO₂ is maintained at a constant 50% throughout the entire surgical procedure. After preoxygenation with 80% FiO₂ for 3 minutes, the FiO₂ is set at 0.50 immediately after intubation and is not modified in response to patient physiology or ORI measurements. PEEP is fixed at 5 cmH₂O, and a standardized alveolar recruitment maneuver is applied at the beginning of surgery. This fixed-FiO₂ strategy differs from the ORI-guided titration group by avoiding dynamic oxygen adjustments and reflects conventional intraoperative oxygen management commonly used in clinical practice.
  Other Names: fixed 50:50 oxygen and air combination
  Arms: Group 2- Fixed FiO₂

SUMMARY:
Atelectasis is a frequent pulmonary complication after general anesthesia, often triggered by preoxygenation and intraoperative hyperoxia. High inspiratory oxygen fractions (FiO₂) can promote absorption atelectasis, ventilation-perfusion mismatch, hemodynamic alterations, and oxidative injury.

This study evaluates the effect of two intraoperative oxygen management strategies-oxygen reserve index (ORI)-guided FiO₂ titration versus fixed 50% FiO₂-on postoperative atelectasis in patients undergoing thoracolumbar spine surgery under general anesthesia. Atelectasis severity will be assessed using lung ultrasonography (LUS), scored across 12 thoracic regions (0-3 per region, total 0-36), while respiratory function changes will be examined via preoperative and 24-hour postoperative spirometry (FVC, FEV₁, FEV₁/FVC).

Because postoperative spirometry may be influenced by pain, Numeric Rating Scale (NRS) scores will be recorded to help distinguish true restrictive patterns from pain-limited respiratory effort.

The study aims to determine whether ORI-guided FiO₂ titration can reduce postoperative atelectasis and improve respiratory outcomes compared with a fixed FiO₂ approach.

DETAILED DESCRIPTION:
Atelectasis is one of the most common pulmonary complications following general anesthesia, and both preoxygenation and intraoperative hyperoxia are major contributing factors. Hyperoxia can lead to absorption atelectasis, ventilation-perfusion mismatch, cerebral and coronary vasoconstriction, decreased cardiac output, and oxidative tissue injury caused by reactive oxygen species. The use of a high inspiratory oxygen fraction (FiO₂) during general anesthesia, particularly in prolonged surgeries, increases the risk of absorption atelectasis.

This study aims to investigate the impact of different intraoperative oxygen management strategies-oxygen reserve index (ORI)-guided FiO₂ titration versus fixed 50% FiO₂-on the development of postoperative atelectasis in patients undergoing thoracolumbar spine surgery under general anesthesia. The presence and severity of atelectasis will be assessed using lung ultrasonography (LUS), and changes in respiratory function will be evaluated objectively through spirometry measurements.

Lung ultrasonography will be performed by the same experienced and certified anesthesia practitioner for both groups. LUS assessment will be conducted in 12 regions (superior and inferior zones along the anterior, lateral, and posterior lines of each hemithorax). Each region will be scored from 0 to 3 according to the degree of aeration:

0 = normal aeration (A-lines predominance, <2 B-lines);

1. = mild loss of aeration (≥3 well-defined B-lines);
2. = moderate loss of aeration (multiple coalescent B-lines or "white lung");
3. = severe loss of aeration (subpleural or complete consolidation with air bronchograms).

The total LUS score ranges from 0 to 36, with higher scores indicating greater loss of aeration and presence of atelectasis.

Spirometry will be performed preoperatively and at 24 hours postoperatively, with patients in a seated position using a nose clip and a single-use cardboard mouthpiece. After a maximal inspiration, patients will be instructed to perform a forceful and sustained expiration according to device guidance. At least three maneuvers will be recorded, and the best values for FVC, FEV₁, and FEV₁/FVC will be documented.

Postoperative spirometry results may be influenced by pain, as inadequate inspiration or shortened expiration can lead to artificially reduced FVC and FEV₁ values. Therefore, postoperative pain will be assessed using the Numeric Rating Scale (NRS, 0-10), enabling differentiation between true atelectasis-related restrictive patterns and pain-limited respiratory effort.

This study focuses on optimizing oxygenation and preventing postoperative pulmonary atelectasis caused by higher intraoperative oxygen exposure in patients undergoing elective thoracolumbar spine surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 80 years
2. Patients with an ASA physical status of I, II, or III
3. Individuals with a body mass index (BMI) between 18 and 35 kg/m²

Exclusion Criteria:

1. History of or active upper or lower respiratory tract infection within the past month
2. Pulmonary emphysematous/bullous disease or COPD
3. Pre-existing significant atelectasis or consolidation (Preoperative LUS showing a score of 3 consolidation or ≥2 regions with a score ≥2)
4. Severe obstructive sleep apnea requiring CPAP therapy
5. NYHA class III-IV heart failure, EF <35%, or severe valvular disease
6. Severe arrhythmia or hemodynamic instability requiring high-dose vasopressors
7. Body mass index (BMI) >35 kg/m²
8. Severe anemia (Hb <9 g/dL) or polycythemia (Hb >18 g/dL)
9. Non-diagnostic or unclear preoperative lung ultrasound images
10. Preoperative SpO₂ ≤ 94%
11. Inability to apply the sensor due to finger deformity, or inadequate signal caused by digital hypoperfusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Total Lung Ultrasound (LUS) Score | Baseline (Preoperative) and 30 Minutes After Extubation
  The primary outcome of the study is the change in the total Lung Ultrasound (LUS) score obtained using a standardized 12-zone lung ultrasound protocol. Each hemithorax was evaluated in six regions-anterior, lateral, and posterior lines, each divided into superior and inferior zones-resulting in a total of 12 assessed areas. Each zone was scored from 0 to 3 based on the degree of aeration, yielding a total score ranging from 0 to 36, with higher scores indicating greater aeration loss and atelectasis. Accordingly, the difference between the preoperative LUS score and the LUS score measured at 30 minutes after extubation was defined as the primary endpoint of the study.

SECONDARY OUTCOMES:
Change in Forced Vital Capacity (FVC) | Baseline (Preoperative) and Postoperative 24th Hour
  Spirometry is performed preoperatively and repeated at 24 hours postoperatively. Forced Vital Capacity (FVC) is defined as the total volume of air that can be forcibly exhaled from the lungs after a maximal inhalation.
Change in Forced Expiratory Volume in 1 Second (FEV1) | Baseline (Preoperative) and Postoperative 24th Hour
  Spirometry is performed preoperatively and repeated at 24 hours postoperatively. FEV1 is defined as the volume of air exhaled during the first second of a forced expiration.
Change in FEV1/FVC Ratio | Baseline (Preoperative) and Postoperative 24th Hour
  Spirometry is performed preoperatively and repeated at 24 hours postoperatively. The ratio is calculated by dividing the Forced Expiratory Volume in 1 Second (FEV1) by the Forced Vital Capacity (FVC). The result is multiplied by 100 and expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Derya Özkan, Professor, Study Director — Ankara Etlik City Hospital

IPD SHARING:
Plan to Share IPD: No